CLINICAL TRIAL: NCT03830632
Title: Effects Of Plyometric Training Program On Speed And Agility In Young Cricketers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zohra Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, WAQAR AHMED AWAN, Associate Professor, Zohra Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ZIHS-Rwp/IRC/001
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Physical Fitness
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training Program (Experimental): The plyometric training group participated in a 6-week training program performing a variety of plyometric exercises designed for the lower extremity , while the control group did not participate in any plyometric exercises. All subjects were instructed not to start any lower extremity strengthening programs during the 6-week period and to only perform activities of normal daily living.
  Interventions: Other: Plyometric Training
- Traditional Training (Active Comparator): AEROBIC TRAINING - A minimum of two low-intensity sessions a week consisting of 1 hour running. .
  SHUTTLE SPRINTS - Placed two cones roughly 25 yards apart. Ask cricketer to sprint as fast as back and forth between the cones 12 times, for a total of six round-trips. ask them to finish in one minute. give rest for up to five minutes, then repeat once or twice.
  Interventions: Other: Traditional Training

INTERVENTIONS:
Other: Plyometric Training
  Arms: Plyometric Training Program
Other: Traditional Training
  Arms: Traditional Training

SUMMARY:
This study was to determine the effects of plyometric training program on speed and agility in young cricketer. There were two groups, one received plyometric training program and other received training training to improve speed and agility in young cricketers

DETAILED DESCRIPTION:
Plyometric training has been an effective method for the improvement of agility, sprinting, and jumping ability and it has also been reported to Improve running economy, joint stability, increased joint awareness and overall proprioception and decrease the severity of knee injuries. In the Plyometric exercise involves starting, stopping, and change of movement directions which contribute to agility development.The athletes use plyometric training techniques in many sports to improve explosive power and body strength. The plyometrics is a rapid stretch of muscle (eccentric) contraction straight away shortening (concentric) contraction in similar muscle tissue

ELIGIBILITY:
Inclusion Criteria:

°The male professional cricketers with age between 14-24 years old from Islamabad were included.

Exclusion Criteria:

° Cricketers not engaged in game from last 1 month.

Ages: 14 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Speed Test (10 meter sprint test) | 8 Weeks
  Speed tests are typically used solely to measure an athlete's linear speed capabilities. More specifically, the 10-metre (m) sprint test is used to measure acceleration. Before the introduction of timing gates, speed tests were typically officiated using stopwatches, though stopwatches are still useful and can be used reliably, the use of timing gates is highly recommended and essential when precision is required.
  As the 10m sprint test measures acceleration from a static position, it is a common testing protocol as a large majority of sports often involve such short-distance sprint movements. Sports that include any form of short-distance acceleration should often include a 10m sprint test in their performance testing battery.
Agility T-Test | 8 Weeks
  the T-Test is a test of agility for athletes, and includes forward, lateral, and backward running. equipment required: tape measure, marking cones, stopwatch, timing gates.
  Test setup: Set out four cones Procedure: The subject starts at cone A. On the command of the timer, the subject sprints to cone B and touches the base of the cone with their right hand. They then turn left and shuffle sideways to cone C, and also touches its base, this time with their left hand. Then shuffling sideways to the right to cone D and touching the base with the right hand. They then shuffle back to cone B touching with the left hand, and run backwards to cone A. The stopwatch is stopped as they pass cone A. Take the best time of three successful trials to the nearest 0.1 seconds.